CLINICAL TRIAL: NCT03597542
Title: Examining the Relationship Between Acute Meal Intake and Inflammation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, Naiman Khan, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17112
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Inflammation
Keywords: Children; Inflammation; Obesity
MeSH Terms: conditions — Obesity; Inflammation | interventions — Eggs; Carbohydrates

STUDY DESIGN:
Intervention Model Description: Double blind randomized cross-over design
Who Masked: Participant, Investigator
Masking Description: Both the participants and researchers involved with data analysis will be blinded to which condition given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maltodextrin (Experimental): Participants will consume 56g of maltodextrin dissolved in 500mL of water.
  Interventions: Other: Eggs and Carbohydrates
- Egg (Experimental): Participants will consume 36g of spray-dried egg powder (equivalent to 3 eggs) dissolved in 500mL of water.
  Interventions: Other: Eggs and Carbohydrates

INTERVENTIONS:
Other: Eggs and Carbohydrates — Participants are asked to consume both egg based powder or maltodextrin dissolved in 500mL of water at two different time points at least one week apart. Participants will then submit to a venous blood draw to assess levels of cellular inflammation.

SUMMARY:
Recent evidence has shown that obese and overweight children exhibit states of chronic inflammation. In obese adults, a high carbohydrate meal induces an inflammatory response; however, the effects of a high carbohydrate meal on biomarkers of inflammation has not previously been examined in children. The purpose of this research project is to characterize the inflammatory response to a high carbohydrate versus a low carbohydrate meal in healthy weight, overweight, and obese children (age 7-17 years). After completing informed consent/assent, a Dual-energy X-ray Absorptiometry (DXA) scan, and baseline blood draw on experimental day 1, children will then return to the lab two times to ingest either a high or low carbohydrate beverage followed by post-meal blood collection for a total of 3 blood draws. Biomarkers of inflammation will be analyzed by flow cytometry and enzyme-linked immunosorbent assay (ELISA). Participants will be recruited through various studies through the Neurocognitive Kinesiology Lab/Body Composition and Nutritional Neuroscience Labs as well as through the local Champaign-Urbana community. Data from this project will provide a better understanding of the inflammatory response to different meals in healthy weight, overweight, and obese children.

ELIGIBILITY:
Inclusion Criteria:

• Between the ages of 7-17

Exclusion Criteria:

* Younger than 7 years and older than 17 years
* Presence of allergies to eggs and/or sugar substitutes
* Presence of heart or respiratory disease
* Presence of uncontrolled hypertension, diabetes
* Use of anti-inflammatory medications
* Presence of cancer or metabolic disease

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Effects of egg or maltodextrin on inflammatory cytokines (Tumor necrosis factor-alpha, C-reactive protein, and Interleukin-6) | 3 weeks.
  Will be used by determining any changes in inflammatory cytokines via enzyme-linked immunosorbent assay (ELISA) kits.

SECONDARY OUTCOMES:
Effects of egg or maltodextrin on inflammatory monocyte cells with and without expression of Toll-like receptor 4 and C-C Chemokine receptor-2. | 3 weeks.
  Will be used by determining the cells per microliter of lysed whole blood.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niemiro GM, Chiarlitti NA, Khan NA, De Lisio M. A Carbohydrate Beverage Reduces Monocytes Expressing TLR4 in Children with Overweight or Obesity. J Nutr. 2020 Mar 1;150(3):616-622. doi: 10.1093/jn/nxz294. PMID 31825075